CLINICAL TRIAL: NCT01152502
Title: Paracetamol Metabolism in Post Operative Conditions
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Patrick LACARIN, CHU Clermont-Ferrand
Other Study IDs: CHU-0076
Record Dates: First submitted 2010-06-28; First posted 2010-06-29 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2010-06

CONDITIONS: Aortic Surgery and Treatment Post Operative With Paracetamol During 4 Days
Keywords: Post operative conditions, paracetamol metabolites

STUDY DESIGN:
Time Perspective: Cross-Sectional

SUMMARY:
Follow-up of urinary concentration from paracetamol metabolites by patients with aortic surgery during 4 days therapeutic intake (perfalgan ® 4 x 1g IV/day)

DETAILED DESCRIPTION:
D-15 to D0: selection

* patient information and non-opposition obtained
* inclusion and non inclusion criteria check
* clinical exam

D-1 to D0 : 24 hours diuresis

D0 : operation day

Before anesthesia :

* urine collection (paracetamol metabolites dosage)
* blood sampling (glutathion and liver function test)

Surgery:

* 1st paracetamol intake before closing
* Then administration every 6 hours

D1 to D4 :

* 24 hours urine collection (metabolites dosage)
* blood sampling et D1 and D4(glutathion and liver function test)

D5 : final clinical exam

ELIGIBILITY:
Inclusion Criteria:

* aortic surgery
* treatment with intraveinous paracetamol (4 grammes daily during 4 days)
* patient agrees to participate

Exclusion Criteria:

* - patient disagrees
* paracetamol contra-indication
* paracetamol intake 5 days before surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Defined population
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2008-06; Primary Completion 2008-09 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Follow-up of urinary concentration from paracetamol metabolites by patients with aortic surgery during 4 days therapeutic intake (perfalgan ® 4 x 1g IV/day) | during 4 days therapeutic intake

SECONDARY OUTCOMES:
- Follow-up of glutathion concentration during 4 post operative days | during 4 post operative days
Monitoring of liver function

CONTACTS AND LOCATIONS:
Overall Officials: Eric SCHNEIDER, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France